CLINICAL TRIAL: NCT04252937
Title: A Dose Escalation Evaluation of Safety and Tolerability of Adrecizumab - a Humanized Monoclonal Antibody Against Adrenomedullin (ADM) in Patients With Acute Heart Failure Requiring Hospitalization
Brief Title: Adrecizumab Dose Escalation Safety and Tolerability Evaluation (ADESTE)
Acronym: ADESTE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GREAT Network Italy (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Adeste Study
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure treatment Adrecizumab Safety
MeSH Terms: interventions — enibarcimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAM8101 (Adrecizumab) : 0.5 mg/kg (Experimental): HAM8101 (Adrecizumab) : 0.5 mg/kg
  Interventions: Drug: Adrecizumab
- HAM8101 (Adrecizumab) : 2 mg/kg (Experimental): HAM8101 (Adrecizumab) : 2 mg/kg
  Interventions: Drug: Adrecizumab
- HAM8101 (Adrecizumab) : 8 mg/kg (Experimental): HAM8101 (Adrecizumab) : 8 mg/kg
  Interventions: Drug: Adrecizumab

INTERVENTIONS:
Drug: Adrecizumab — HAM8101 (Adrecizumab) is a humanized IgG1 monoclonal antibody (mAb).
  Other Names: HAM8101 (Adrecizumab)

SUMMARY:
This is an open, standard therapy controlled clinical trial using a single intravenous infusion of HAM8101 (Adrecizumab) in patients hospitalized for AHF. This study will serve as a safety trial for HAM8101 (Adrecizumab) in AHF, using a dose escalating design.

Acute Heart Failure (AHF), both as deterioration of chronic stable condition or "de novo" onset constitutes a major indication of particular interest and continues to be a major health problem, with millions of people being affected, still associated with high mortality and rehospitalization rates despite numerous attempts to improve the situation.

It is believed that deteriorated vascular integrity and function, which manifests in various symptoms resulting from extravasation of fluid and solutes, is a key mechanism contributing to development and progression of the disease.

Therefore, it is warranted to start a phase 2 safety and proof of concept study with a new investigational product (IMP) that enhances the plasma concentration of bio-ADM in the circulation to restore and stabilize the vascular integrity and function in patients with AHF after initial stabilization with the current standard of care (SoC).

DETAILED DESCRIPTION:
The objectives of this study are to determine the safety/tolerability together with PD parameters of an intravenous slow infusion of 3 increasing doses of HAM8101 (Adrecizumab) in patients with AHF in a Phase IIa safety clinical trial. Efficacy of HAM8101 (Adrecizumab) will be explored secondarily.

The primary objective of this trial is to evaluate safety and tolerability of increasing doses of HAM8101 (Adrecizumab) in patients with AHF. Treatment emergent SAEs will be collected and carefully monitored on a continuous basis during the in-hospital stay and the 3-month follow-up after discharge. Treatment emergent AEs will be collected and monitored on a continuous basis during the in-hospital stay. Plasma and urine specimens will be collected daily from the first day of treatment until hospital discharge for routine safety assessments and to evaluate renal function.

All subjects will receive phone calls 30 (±7) days from start of study drug infusion to assess the occurrence of adverse events and serious adverse events, mortality and hospital readmission for HF or renal dysfunction. Patients will be contacted again 60 (±14) days and 90 (±14) days after infusion of HAM8101 (Adrecizumab) to document survival and episodes of re-hospitalization.

The study is designed primarily to understand the safety and tolerability of increasing doses of HAM8101 (Adrecizumab) in AHF patients (NYHA class II-IV) already in treatment and hemodynamically stabilized with a therapy that represents the standard of care (SoC) as recommended by international ESC 2016 Guidelines and it comprises 3 different patient "cohorts" with each cohort receiving one of 3 escalating doses of HAM8101 (Adrecizumab).

In addition, the study will provide a PD profile of HAM8101 (Adrecizumab) in AHF, in this acute condition.

After signing an Institutional Review Board approved Informed Consent Form, subjects will be asked to undergo screening procedures for study eligibility. Patients will be prescreened by site staff based on potential entry criteria as soon as possible after admission. Upon confirmation of eligibility and informed consent signature, the patient will receive the study drug within 48h from hospital admission. All patients will be evaluated daily during the hospitalization. In-hospital assessments of symptoms and signs of residual congestion (as composite congestion score) will be made daily from start of study drug infusion and up to Day 7, unless a patient is discharged earlier or later or dies earlier than Day 7. After discharge patients will be followed up for an additional 3 months for safety assessments with telephone contacts at months 1, 2, and 3, to document survival and episodes of re-hospitalization.

Thirty (30) patients with AHF (NYHA class II-IV) will be enrolled into 3 sequential experimental cohorts during the inpatient setting: 0.5 mg/kg, 2 mg/kg and 8 mg/kg of HAM8101 (Adrecizumab).

A control group of 10 patients with AHF will receive only standard of care treatment and will be monitored during the inpatient and outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Hospitalization due to the primary diagnosis of AHF, based on ESC 2016 Guidelines;
3. NYHA II/III/IV;
4. Must be able to be enrolled within 48h from admission to the hospital;
5. Body weight 50 - 120 kg;
6. Able and willing to provide informed written consent and written documentation of informed consent.

Exclusion Criteria:

1. NYHA Class I;
2. Dyspnea primarily due to non-cardiac causes;
3. Clinical diagnosis of acute coronary syndrome, planned PCI, life-threatening arrhythmias, planned ICD/CRT, planned cardiac surgery;
4. Recent CABG and PCI in the last 3 months;
5. Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy, congenital disease, uncorrected primary valve disease needing cardiac surgery;
6. Ongoing or planned treatment with ultrafiltration or dialysis;
7. Patients that required cardiopulmonary resuscitation in the last 4 weeks prior to enrollment;
8. Systolic blood pressure at enrolment <100 mmHg or >180 mmHg;
9. Current (within 2h prior to screening) need of cardiac/respiratory mechanical support;
10. Severe pulmonary disease with chronic oxygen need at home or history of COPD >GOLD III, IPF or Bronchial Asthma;
11. Any condition or therapy, which would make the patient unsuitable for the study, or life expectancy less than 12 months (e.g. active malignancy);
12. Impaired renal function with eGFR <30 ml/min/1.73 m² calculated by Modification of Diet in Renal Disease [MDRD] formula;
13. Anemia (Hb <9 g/L or hematocrit <25%);
14. Temperature >38°C (oral or equivalent) or sepsis or active infection requiring IV antimicrobial treatment;
15. Hepatic insufficiency classified as Child-Pugh B or C;
16. Any organ transplant recipient, or patient currently listed for transplant or admitted for any transplantation;
17. Major surgery within 30 days;
18. Unwilling or unable to be fully evaluated for all follow-up assessments;
19. Participation in an interventional clinical trial involving another investigational drug or an implantable medical device within 4 weeks prior to inclusion;
20. Women of child bearing potential or women who are pregnant or breast-feeding or are not using adequate contraceptive methods [i.e. orally administered hormonal contraceptives, surgical intervention (tubal ligation), intrauterine device (IUD) and sexual abstinence];
21. Male patients with reproductive potential who refuse adequate means of contraception during and up to 3 months after end of infusion of HAM8101 (Adrecizumab).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Serious Adverse Events (SAEs) during the hospitalization period | 7 days

SECONDARY OUTCOMES:
In-hospital assessment of AHF | 7 days
  Change in signs and symptoms of AHF assessed at 30min, 1h, 6h, 12h, 24h from onset of test dose and daily through day 7 - or until discharge from hospital if this occurs earlier or later than 7 days. For "change" is intended a change in severity of considered signs and symptoms (e.g. shift from moderate to mild or vice versa, etc) symptoms (such as breathlessness, ankle swelling, and fatigue) and signs (e.g. raised jugular venous pressure, pulmonary crackles, peripheral edema, heart gallop sounds and or murmurs, oliguria)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Di Somma, Study Director — GREAT Network Italy
Locations (2):
- Indonesia (2):
  - RSUD Dr. Saiful Anwar Malang, Malang
  - Faculty of Medicine, Public Health and Nursing Universitas Gadjah Mada, Yogyakarta

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available

REFERENCES:
- [Background] Geven C, Pickkers P. The mechanism of action of the adrenomedullin-binding antibody adrecizumab. Crit Care. 2018 Jun 13;22(1):159. doi: 10.1186/s13054-018-2074-1. No abstract available. PMID 29895302
- [Background] Geven C, van Lier D, Blet A, Peelen R, Ten Elzen B, Mebazaa A, Kox M, Pickkers P. Safety, tolerability and pharmacokinetics/pharmacodynamics of the adrenomedullin antibody adrecizumab in a first-in-human study and during experimental human endotoxaemia in healthy subjects. Br J Clin Pharmacol. 2018 Sep;84(9):2129-2141. doi: 10.1111/bcp.13655. Epub 2018 Jul 3. PMID 29856470
- [Background] Ambrosy AP, Pang PS, Khan S, Konstam MA, Fonarow GC, Traver B, Maggioni AP, Cook T, Swedberg K, Burnett JC Jr, Grinfeld L, Udelson JE, Zannad F, Gheorghiade M; EVEREST Trial Investigators. Clinical course and predictive value of congestion during hospitalization in patients admitted for worsening signs and symptoms of heart failure with reduced ejection fraction: findings from the EVEREST trial. Eur Heart J. 2013 Mar;34(11):835-43. doi: 10.1093/eurheartj/ehs444. Epub 2013 Jan 4. PMID 23293303